CLINICAL TRIAL: NCT04861740
Title: Autism Access Link for Early Referral and Treatment
Acronym: Autism ALERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Boston Medical Center (Other); Providence Health & Services (Other)
Responsible Party: Principal Investigator, Katharine Zuckerman, MD MPH, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 00001
Record Dates: First submitted 2021-04-07; First posted 2021-04-27 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Primary Care; Case Management
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Mass Screening

STUDY DESIGN:
Intervention Model Description: We propose a pilot clustered interventional trial with two arms. Clinics in the intervention arm (Screening + Autism ALERT) receive Autism ALERT plus an ASD screening intervention, and clinics in the comparison intervention arm (Screening Only) receive the ASD screening intervention only (START Autism). As this is a pilot trial, primary outcomes of interest are feasibility and acceptability. We will additionally assess mechanism of outcome, preliminary efficacy, and protocol fidelity. Feasibility and acceptability will be assessed in intervention clinics. Mechanism of action and preliminary efficacy will be assessed by comparing intervention to control clinics. Fidelity is assessed in both arms. We will pilot test Autism ALERT in 6 safety-net primary care clinics in Oregon.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Screening + Autism ALERT (Experimental): Clinics in the intervention arm receive Autism ALERT plus an ASD screening intervention (START Autism).
  Interventions: Other: Autism ALERT; Other: Screening Intervention
- Screening Only (Active Comparator): Clinics in the comparison intervention (control) arm receive the ASD screening intervention only (START Autism).
  Interventions: Other: Screening Intervention

INTERVENTIONS:
Other: Autism ALERT — Autism Access Link for Early Referral and Treatment [ALERT], the intervention proposed in this application, is a novel state-wide referral and case management platform that PCPs can activate to ensure that a child with suspected ASD receives all necessary ASD diagnosis and treatment resources in a single referral, radically simplifying a complex diagnostic and treatment process.
  Arms: Screening + Autism ALERT
Other: Screening Intervention — Autism screening intervention only.
  Other Names: START Autism

SUMMARY:
Autism Access Link for Early Referral and Treatment [ALERT], the intervention proposed in this application, is a novel state-wide referral and case management platform that PCPs can activate to ensure that a child with suspected ASD receives all necessary ASD diagnosis and treatment resources in a single referral, radically simplifying a complex diagnostic and treatment process. We hypothesize that Autism ALERT will have strong acceptability and high rates of use among primary care providers as well as among diverse low-income patients of children at risk for ASD, and that we will see higher rates of child ASD educational evaluations within six months, and shorter time between referral and ASD treatment, compared with our control.

DETAILED DESCRIPTION:
Though significant research effort has focused on autism spectrum disorder (ASD) screening, less attention has been devoted to optimizing follow-up of children who are subsequently identified as at-risk. Despite increases in ASD screening rates, many children with ASD wait years between when autism is suspected in the primary care setting and when definitive diagnosis and treatment begin. Delayed and missed diagnoses are particularly problematic for low-income and racial/ethnic minority children in the US, who experience higher rates of these adverse outcomes. In this project, we propose to pilot test Autism Access Link to Early Referral and Treatment (Autism ALERT), a statewide monitoring and case management program to accelerate access to ASD diagnosis and treatment among children with suspected ASD the primary care setting. The system will reduce the time between identification of suspected ASD in the primary care setting and establishment of ASD diagnosis and treatment services, by reducing family barriers to care, decreasing primary care provider burdens, and simplifying referral processes. The program will be available to any Oregon child age 12-54 months, regardless of health system or payor type. Autism ALERT will become part of the Help Me Grow national network, which gives it potential for statewide and national spread. In this proposed research, we will pilot test Autism ALERT by comparing it to an existing ASD screening intervention in 6 Oregon primary care practices. Primary goals of this pilot project are to assess feasibility and acceptability of Autism ALERT for primary care providers and families, to test the mechanism of action of Autism ALERT, to pilot test efficacy in reducing time to autism diagnosis and treatment, and to test fidelity of protocol implementation. If successful, this project will be expanded into an implementation/effectiveness R01 in which the program will be tested throughout the state of Oregon. In the long term, this research will result in a sustainable, evidence-based statewide and ultimately national monitoring system children with suspected ASD.

ELIGIBILITY:
Inclusion Criteria:

child's primary care provider suspects the child has ASD, child is patient at one of the study clinics, child age 12 to 54 months, family speaks English or Spanish, no prior ASD medical diagnosis or ASD diagnostic evaluation

Exclusion Criteria:

Previous diagnosis of ASD or prior diagnostic evaluation for ASD.

Ages: 12 Months to 54 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Change in satisfaction with Care Coordination in general and for autism in particular | At enrollment and study end (~9 months after enrollment)
  2 separate provider survey measures
Change in Parent stress | At enrollment and 6 months after enrollment
  Parent Survey - Parenting Stress Index
Change in Parenting stress | At enrollment and 6 months after enrollment
  Questionnaire on Resources and stress - Short Form
Change in Family Empowerment | At enrollment and 6 months after enrollment
  Parent Survey - Family Empowerment Scale, Family Subscale
Change in Family Centered and Coordinated Care | At enrollment and 6 months after enrollment
  Parent Survey - Items from National Survey of Children's Health, Medical Home item set
Family Satisfaction with Program | 6 months after enrollment - Autism ALERT + Screening arm only
  Parent Survey items - Satisfaction with Interpersonal Relationship with Navigator (PSN-I), Client Satisfaction Questionnaire - 8
% referred to program who complete an ASD educational evaluation within 6 months | 6 months after enrollment
  Administrative data - Oregon Early Intervention/Early Childhood Special Ed (EI/ECSE) database
Time from EI/ECSE referral to ASD treatment in EI/ECSE, among children with ASD | measured 9 months after enrollment
  Administrative data - Oregon EI/ECSE database
Family self-reported ASD knowledge | At enrollment and 9 months after enrollment
  5-item survey measure
Change in provider self-efficacy about autism management | At enrollment and at study end (~9 months after enrollment)
  1-item survey measure

SECONDARY OUTCOMES:
Change in provider autism paperwork burden | At enrollment and at study end (~9 months after enrollment)
  Provider survey item
Time from EI/ECSE referral to evaluation among children with ASD | measured 9 months after enrollment
  Administrative data - Oregon EI/ECSE database
Age of EI/ECSE educational determination, among children with ASD | measured 9 months after enrollment
  Administrative data - Oregon EI/ECSE database
% with ASD determination receiving ASD services 6 months after enrollment | measured 9 months after enrollment
  Administrative data - Oregon EI/ECSE database
monthly service hours among children with ASD 6 months after enrollment | measured 9 months after enrollment
  Administrative data - Oregon EI/ECSE database
age of ASD medical diagnosis among children on Medicaid | Measured 1 year after study enrollment
  Administrative data - Medicaid claims
% with ASD medical diagnosis receiving ASD therapy 6 months after enrollment, among children on Medicaid | Measured 1 year after study enrollment
  Administrative data - Medicaid claims

CONTACTS AND LOCATIONS:
Locations (1):
- Ohsu Cdrc, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share data through the NIMH Data Archive as required by the grant.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available indefinitely starting with the conclusion of the study.

REFERENCES:
- [Derived] Zuckerman KE, Owens Reinitz M, Solgi M, Feryn A, Tae M, Cavanaugh P, Raja-Vora J, Fombonne E. Preliminary Efficacy of Telehealth Family Navigation for Early Autism Services Access. J Autism Dev Disord. 2025 Dec 29. doi: 10.1007/s10803-025-07189-w. Online ahead of print. PMID 41460569